CLINICAL TRIAL: NCT06970405
Title: Randomized, Double-Blind, Placebo-Controlled Study of Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Effects of Garetosmab in Men and Post-Menopausal Women With Obesity Who Are Otherwise Healthy
Brief Title: Study of Safety and Effects of Garetosmab in Healthy Obese Men and Post-Menopausal Women
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R2477-OB-2470
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: Healthy; Postmenopausal
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose (Experimental): Randomized per the protocol
  Interventions: Drug: Garetosmab
- Low Dose (Experimental): Randomized per the protocol
  Interventions: Drug: Garetosmab
- Placebo (Placebo Comparator): Randomized per the protocol
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Garetosmab — Administered per the protocol
  Other Names: REGN2477
  Arms: High Dose; Low Dose
Drug: Matching Placebo — Administered per the protocol
  Arms: Placebo

SUMMARY:
This study is researching an experimental drug called garetosmab, referred to as "study drug". The study is focused on otherwise healthy participants with obesity.

The aim of the study is to see how safe and tolerable the study drug is.

The study is looking at several other research questions, including:

* How much study drug is in the blood at different times
* What effect the study drug has on the blood clotting
* What effect the study drug has on hormone levels
* What effect the study drug has on some organs that produce hormones
* What effect hormones have on the side effects produced by the study drug
* Whether the body makes antibodies against the study drug (which could change how well the drug works or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants with obesity (defined as Body Mass Index (BMI) ≥30 kg/m2) who are otherwise healthy, as defined in the protocol
2. Women must be postmenopausal, as defined in the protocol
3. Serum testosterone within age-adjusted normal range for men at screening
4. The platelet count is within the normal lower and upper laboratory range

Key Exclusion Criteria:

1. Patients diagnosed with Type 1 or Type 2 diabetes, as defined in the protocol
2. History of any severe, non-traumatic bleeding, and or a known pre-existing medical history of a bleeding, as defined in the protocol
3. History of clinically significant cardiovascular (eg, uncontrolled blood pressure), endocrine, respiratory, hepatic, renal, gastrointestinal, hematological, psychiatric, or neurological disease, as defined in the protocol
4. Any malignancy in the last 5 years prior to screening visit, except for non-melanoma skin cancer that have been resected with no evidence of metastatic disease
5. Any chronic active infection or has received anti-Hepatitis C Virus (HCV) treatments within the previous 6 months, as defined in the protocol
6. Antiplatelet therapy (eg clopidogrel, aspirin), anticoagulants (eg, warfarin, heparin, factor Xa inhibitor, or thrombin inhibitors) in the last 90 days or within 5 half-lives of the therapy at screening, whichever is longer
7. Use in the previous 90 days for >7 consecutive days at screening of anti-obesity medications, anabolic agents, systemic steroids, androgens, estrogens, or progestogens. Chronic stable doses of thyroid hormones in participants with normal thyroid function are allowed
8. For women, current use, or past use in the last 90 days at screening of hormonal replacement or contraceptive therapy

NOTE: Other Protocol-defined Inclusion/Exclusion Criteria Apply

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05-29 (Estimated); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Through Week 32
Severity of TEAEs | Through Week 32

SECONDARY OUTCOMES:
Change in serum Follicle Stimulating Hormone (FSH) level in response to gonadotropin-releasing hormone (GnRH) injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Percent change in serum FSH level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Change in serum Luteinizing Hormone (LH) level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Percent change in serum LH level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Change in serum total testosterone level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Percent change in serum total testosterone level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Change in serum free testosterone level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Percent change in serum free testosterone level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Change in serum estradiol level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Percent change in serum estradiol level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Change in serum 17-hydroxyprogesterone (17-OHP) level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Percent change in serum 17-OHP level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Change in serum Dehydroepiandrosterone Sulphate (DHEA-S) level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Percent change in serum DHEA-S level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Change in serum androstenedione level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Percent change in serum androstenedione level in response to GnRH injection | Pre-GnRH Baseline, Through Week 20 Post-GnRH
Change in cortisol level in response to Adrenocorticotropic Hormone (ACTH) level injection | Pre-ACTH Baseline, Through Week 20 post-ACTH
Percent change in cortisol level in response to ACTH injection | Pre-ACTH Baseline, Through Week 20 post-ACTH
Concentrations of garetosmab in serum | Through Week 32
Concentrations of total activin A in serum | Through Week 32
Change in bleeding time | Baseline, At Week 8
Percent change in bleeding time | Baseline, At Week 8
Change in thrombin time | Baseline, At Week 8
Percent change in thrombin time | Baseline, At Week 8
Change in Activated Partial Thromboplastin Time (aPTT) | Baseline, At Week 8
Percent change in aPTT | Baseline, At Week 8
Change in Prothrombin Time (PT) | Baseline, At Week 8
Percent change in PT | Baseline, At Week 8
Change in International Normalized Ratio (INR) | Baseline, At Week 8
Percent change in INR | Baseline, At Week 8
Change in platelets count | Baseline, At Week 8
Percent change in platelets count | Baseline, At Week 8
Change in serum ACTH level | Baseline, Through Week 20
Percent change in serum ACTH level | Baseline, Through Week 20
Change in serum FSH level | Baseline, Through Week 20
Percent change in serum FSH level | Baseline, Through Week 20
Change in serum LH level | Baseline, Through Week 20
Percent change in serum LH level | Baseline, Through Week 20
Change in serum Thyroid Stimulating Hormone (TSH) level | Baseline, Through Week 20
Percent change in serum TSH level | Baseline, Through Week 20
Change in serum Thyroxine (T4) level | Baseline, Through Week 20
Percent change in serum T4 level | Baseline, Through Week 20
Change in serum total testosterone level | Baseline, Through Week 20
Percent change in serum total testosterone level | Baseline, Through Week 20
Change in serum free testosterone level | Baseline, Through Week 20
Percent change in serum free testosterone level | Baseline, Through Week 20
Change in serum 17-OHP level | Baseline, Through Week 20
Percent change in serum 17-OHP level | Baseline, Through Week 20
Change in serum estradiol level | Baseline, Through Week 20
Percent change in serum estradiol level | Baseline, Through Week 20
Change in serum DHEA-S level | Baseline, Through Week 20
Percent change in serum DHEA-S level | Baseline, Through Week 20
Change in serum androstenedione level | Baseline, Through Week 20
Percent change in serum androstenedione level | Baseline, Through Week 20
Change in serum Human Growth Hormone (HGH) level | Baseline, Through Week 20
Percent change in serum HGH level | Baseline, Through Week 20
Change in serum Insulin-like Growth Factor (IGF)-1 level | Baseline, Through Week 20
Percent change in serum IGF-1 level | Baseline, Through Week 20
Change in serum cortisol level | Baseline, Through Week 20
Percent change in serum cortisol level | Baseline, Through Week 20
Incidence of Anti-Drug Antibodies (ADA) to garetosmab | Through Week 32
Titer of ADA to garetosmab | Through Week 32

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/